CLINICAL TRIAL: NCT00063401
Title: A Phase II Study of Cetuximab (C225)/Paclitaxel/Carboplatin for the Initial Treatment of Advanced Stage Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Brief Title: Phase II Study in Patients With Epidermal Growth Factor Receptor (EGFR) + Advanced Stage Ovarian, Primary Peritoneal and Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-009; NCT00070044 (obsolete NCT alias)
Record Dates: First submitted 2003-06-25; First posted 2003-06-27 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Ovarian Cancer; Peritoneal Neoplasms; Fallopian Tube Neoplasms
Keywords: ovarian; primary peritoneal cancer; fallopian tube cancer
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms | interventions — Cetuximab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cetuximab 400 mg/m2 IV (over 120 minutes) on Day 1 of Cycle 1, followed by weekly maintenance doses of 250 mg/m2 IV (over 60 minutes). Paclitaxel 175 mg/m2 IC (over 3 hours) and carboplatin AUC of 6 IV (over 30 minutes) on Day 1 of each cycle. For eligible subjects, maintenance therapy will consist of cetuximab 250 mg/m2/week for up to 6 months.
  Interventions: Biological: Cetuximab:; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Cetuximab: — 400 mg/m2 loading dose, 250 mg/m2 weekly, six 21-day cycles
  Other Names: Erbitux
Drug: Paclitaxel — 175 mg/m2 Day 1, six 21-day cycles
Drug: Carboplatin — AUC = 6 Day1, six 21-day cycles

SUMMARY:
The purpose of this study is to determine the progression-free survival obtained with cetuximab (C225)/paclitaxel/carboplatin in subjects with newly diagnosed advanced stage ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
The population being studied in this trial is subjects with advanced stage ovarian, primary peritoneal and fallopian tube cancer will be enrolled. By receiving combination therapy with cetuximab (C225)/paclitaxel/carboplatin, these subjects will experience longer progression-free survival than previously reported for subjects receiving only paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must have signed an approved informed consent.
2. Subjects with histologic diagnosis of epithelial ovarian carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma, Stage III or IV, with either optimal (≤ 1 cm residual disease) or suboptimal residual disease following initial surgery. All subjects must have had appropriate surgery for ovarian, primary peritoneal, or fallopian tube carcinoma with appropriate tissue available for histologic evaluation. Pathology must be verified at the participating institution
3. Subjects with the following histologic epithelial cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma N.O.S.
4. Subjects with tumor tissue available for assessment of EGFR status by IHC.
5. EGFR expression must be positive (e.g., 1+).
6. Subjects must have a Karnofsky Performance Status (KPS) of ≥ 70%.
7. Subjects must be entered no more than 12 weeks postoperatively.
8. Women, ages 18 and older.
9. Bone marrow function: absolute neutrophil count (ANC) ≥ 1,500/ul, equivalent to Common Toxicity Criteria (CTC) grade 1. Platelets ≥ the institutional lower limit of normal (LLN), CTC grade 0.
10. Renal function: creatinine ≤ 1.5 x institutional upper limit of normal (ULN), CTC grade 1.
11. Hepatic function: bilirubin ≤ 1.5 x ULN, CTC grade 1. AST ≤ 2.5 x ULN, CTC grade 1.
12. Neurologic function: neuropathy (sensory) ≤ CTC grade 1.

Exclusion Criteria

1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study.
2. WOCBP using a prohibited contraceptive method.
3. Women who are pregnant or breastfeeding
4. Women with a positive pregnancy test on enrollment or prior to study drug administration.
5. Subjects with a current diagnosis of epithelial ovarian tumor of low malignant potential (borderline carcinomas) are not eligible. Subjects with a prior diagnosis of a low malignant potential tumor that was surgically resected and who subsequently develop invasive adenocarcinoma are eligible, provided that they have not received prior chemotherapy for any ovarian tumor.
6. Subjects who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than 3 years prior to registration, and the subject remains free of recurrent or metastatic disease.
7. Subjects who have received prior chemotherapy for any abdominal or pelvic tumor are excluded. Subjects may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than 3 years prior to registration,and that the subject remains free of recurrent or metastatic disease.
8. With the exception of non-melanoma skin cancer and other specific malignancies as noted above, subjects with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy are excluded.
9. Subjects with acute hepatitis.
10. Subjects with active or uncontrolled infection are not eligible.
11. Subjects with a significant history of cardiac disease, i.e., uncontrolled hypertension,unstable angina, and congestive heart failure.
12. Subjects with left ventricular ejection fraction (LVEF) below the institutional range of normal on a baseline multiple gated acquisition (MUGA) scan or echocardiogram.
13. A history of prior cetuximab or other therapy which targets the EGFR pathway or a history of prior chimerized or murine monoclonal antibody therapy.
14. Subjects with a known allergy to murine proteins or Cremophor EL.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To determine the progression-free survival obtained with cetuximab (C225)/paclitaxel/carboplatin in subjects with newly diagnosed advanced stage ovarian, primary peritoneal, or fallopian tube cancer. | How long patients have progression-free survival

SECONDARY OUTCOMES:
To determine clinical and/or pathological response rates with cetuximab (C225)/paclitaxel/carboplatin in subjects with newly diagnosed advanced stage ovarian, primary peritoneal, or fallopian tube cancer. | Length of time for a response to treatment
To evaluate the toxicity of the combination regimen in this subject population. | Length of time for a response to treatment
To access EGFR expression by immunohistochemical assay. | Length of time for a response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Philadelphia, Pennsylvania